CLINICAL TRIAL: NCT05419661
Title: Evaluation of the Interest of a Simulated Procedure Performed on a Printed Model in the Endovascular Treatment of Carotid-sylvian Aneurysms
Brief Title: Interest of a Simulated Procedure Performed on a Printed Model in the Endovascular Treatment of Carotid-sylvian Aneurysms
Acronym: Anev3D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 29BRC20.0132
Record Dates: First submitted 2022-05-23; First posted 2022-06-15 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Aneurysm Cerebral
Keywords: Operational Pre-Planning; embolization; 3D printer; carotid-sylvian aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPO + (Experimental): Operational Pre-Planning + intracranial aneurysm embolization treatment
  Interventions: Other: Operational Pre-Planning
- PPO - (No Intervention): Only intracranial aneurysm embolization treatment

INTERVENTIONS:
Other: Operational Pre-Planning — Using a 3D printer, printing of the patient's aneurysm from the segmented 3D images obtained during the initial assessment and thus allowing a simulation of the embolization procedure. This pre-operative planning (PPO) carried out in real conditions aims to anticipate the possible complications that could be encountered on the same day of treatment.
  Other Names: PPO
  Arms: PPO +

SUMMARY:
It is now considered that 1% to 2% of the French population has an intracranial aneurysm. The major risk of this malformation is essentially the rupture which will lead in 10% of cases to death immediately, in 30% to 50% death within three weeks and in 30% of cases the patients will present a permanent disability. The management of this pathology represents today a major health challenge. Historically, neurosurgery was the discipline of first choice for the treatment of this pathology. This consists of clipping the aneurysm by a surgical approach to exclude it from the blood circulation and thus avoid its rupture. For many years now, interventional neuroradiology has established itself, through its "minimally invasive" and endovascular approach, as the reference treatment for ruptured and non-ruptured intracranial aneurysms: this is embolization. This so-called minimally invasive technique consists of placing directly into the aneurysm, using micro-catheters that are navigated under radiological control from the femoral artery, turns of plates called "coils" or prostheses called " stent" or "flow-diverter". This technique makes it possible to secure the aneurysm from the inside and thus reduce the risk of rupture. Today, 95% of patients are treated using this innovative technique and limited intraoperative risks. Interventional neuroradiology has constantly known in recent years a set of revolutions and innovations in terms of implantable medical devices (IMD) allowing to treat more and more patients with excellent clinical results. Today, the interventional neuroradiologist, assisted by the radiographer, has a very wide range of IMDs that he can combine with each other depending on the type, location, size and shape of the aneurysm. The role of the manipulator, here, is to work closely with the neuroradiologist so that he has, on the one hand, quality images and on the other hand, that he can count on a precious ally, an expert in IMDs, during embolization procedures. However, the wide choice of medical devices and the complexity of the aneurysms to be treated sometimes make treatment complicated. On the day of the "cold" treatment of the aneurysm (i.e. non-ruptured), the technicality of the catheterization and aneurysm's spatial conformation complicates the deployment of embolization equipment. This then sometimes leads to undesirable events such as intraoperative rupture. The very purpose of this study is to be able, by means of a 3D printer, to print the patient's aneurysm from the segmented 3D images obtained during the initial assessment and thus proceed to a simulation of the embolization procedure. This pre-operative planning (PPO) carried out in real conditions aims to anticipate the possible complications that could be encountered on the same day of treatment.

DETAILED DESCRIPTION:
The indication of a primary preventive treatment by endovascular route will be posed in a multidisciplinary consultation meeting of neurovascular pathology for patients who have accidentally discovered a carotid-sylvian cerebral aneurysm (not ruptured).

During the treatment announcement consultation carried out by an interventional neuroradiologist taking place, generally less than a month, after the staff, the latter may propose the study to the patient. The investigator gives him the information letter. The patient will benefit from a reflection period of one week and will be contacted by telephone by the MERM to validate or not his wish to participate in the study.

The random selection of patients is carried out in consultation during the inclusion visit (consultation with the MERM). The pre-operative course will be carried out according to the usual scheme in the 2 groups. Unlike the control group (PPO-), the PPO+ group will have a parallel PPO (Pre-Planning Operative). The intracranial aneurysm embolization treatment procedure will then be performed in both groups.

The duration of the study is a maximum of 6 months per participant, including a maximum interval of 2 months between the inclusion visit and the treatment (usual coverage period between the treatment announcement consultation and the intervention) and 4 months of follow-up (end-of-study visit at M4).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Social security affiliation
* Patient who signed inform consent form
* Patient with an unruptured saccular carotid-sylvian aneurysm of more than 4 mm in long axis and less than 20 mm
* Primary preventive treatment decision validated in CPR
* Patient having benefited from a 3DRA during a previous arteriography dating from less than 6 months, or whose cerebral arteriography is planned less than 2 weeks before the intervention

Exclusion Criteria:

* Unable or unwilling to come for follow-up appointments
* Weight > 250kg due to weight limits on the angiographic table
* Allergy to iodinated contrast agents
* Patient with a contraindication to MRI
* Pregnancy, breastfeeding or planning to become pregnant in the following year
* Limited life expectancy < 1 year
* Patient participating in another clinical study or having completed their participation less than 30 days ago
* Patient under legal protection, Patient under guardianship or curatorship
* Kidney failure, GFR < 60ml/min/1.73 m2
* Platelets < 50 x 10 ^ 9/L
* Partially thrombosed aneurysm
* Partially calcified aneurysm
* Recanalized or previously treated aneurysm (coils, stent, clip, flow disrupter)
* Another aneurysm on the same carrier artery already treated (coils, stent, clip, flow disrupter)
* Ruptured aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Failure rate during implantation of the first two implantable devices chosen, failure being defined as non-implantation of one of the first two implantable devices used. | 15 months

SECONDARY OUTCOMES:
Number of attempts to implant a device | 15 months
device usage time | 15 months
  Catheterization's time and implantation's time
Operative time | 15 months
  time between placement of intermediate catheters in the internal carotid artery and final control
Quantity of X-radiation | 15 months
Quantity of iodinated contrast product | 15 months
General anesthesia time | 15 months
Number of per-procedure adverse events | 15 months
Number of complications related to the procedure | 15 months

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.